CLINICAL TRIAL: NCT04820465
Title: Identification of the Main Causes of Anemia in Older Adults
Brief Title: Anemia in Older Adults
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Principal Investigator, Vanessa De la Cruz, Researcher in Medical Science Level D, Instituto Nacional de Salud Publica, Mexico
Other Study IDs: S0008-2014-1 - 000000000234157
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Anemia; Nutritional Deficiency; Inflammation
Keywords: Anemia; Older mexican adults; Vitamin A deficiency; Iron deficiency; Vitamin B12 deficiency
MeSH Terms: conditions — Anemia; Malnutrition; Inflammation; Vitamin A Deficiency; Iron Deficiencies; Vitamin B 12 Deficiency

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non available due to cross-sectional study design — Non available since this study (survey) has a cross-sectional design

SUMMARY:
A cross-sectional study with 829 older Mexican adults were recruited from July to September 2015, from four localities in the southern region of México. Older adults were interviewed at their homes and a fasting blood sample was obtained for analysis of micronutrient status (iron deficiency, vitamin B12 deficiency, folate deficiency, vitamin A deficiency and biomarkers of inflammation). The aim of the study was to identify the main causes of anemia in older adults with higher rates of anemia according to the recent data of the Mexican National Health and Nutrition Survey.

DETAILED DESCRIPTION:
A survey with cross-sectional design was applied in 829 older Mexican adults, recruited during the period July to September 2015, from four localities in the southern region of México: including Champotón, Campeche, Mérida, and Valladolid. Older adults were interviewed at their homes to collect nutrition, health, cognitive and dietary information. Anthropometric measures and functionallity tests were also collected. A finger prick capillary blood sample was collected to measure hemoblobin in situ using HemoCue. Anemia was defined according to WHO criteria. A fasting venous blood sample was collected in 803 older adults. Serum was separated and frozen at -20°C to measure ferritin, retinol, vitamin B12, folate, iron, soluble transferrin receptor, C-reactive protein, interleukin 6, alpha glycoprotein 1, hepcidin, erythropoietin in the laboratory of nutrition of the National Institute of Public Health.

The study protocol was approved by Research, Biosecurity and Ethics Committees of the National Institute of Public Health. Participants received a detailed explanation of the study procedures and signed an informed consent form prior to data collection.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults who wish to participate in the study
* Ambulatory older adultos
* Older adult with own decision making

Exclusion Criteria:

* Non demented
* Non oxygen dependent
* No disability

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults >=60 years living in urban localities from the southern region of Mexico ( Champotón, Valladolid, Campeche and Yucatán) were visited at their homes. 60% of the total sample were women and the rest men.
Sampling Method: Probability Sample
Enrollment: 829 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Anemia | July- September 2015
  Hemoglobin measure in capillary blood sample

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez RP, De la Cruz-Gongora V, Rodriguez AS. Serum retinol levels are associated with cognitive function among community-dwelling older Mexican adults. Nutr Neurosci. 2022 Sep;25(9):1881-1888. doi: 10.1080/1028415X.2021.1913315. Epub 2021 Apr 13. PMID 33847257